CLINICAL TRIAL: NCT03868683
Title: The Glycemic Effect of Added Sugar on Bake Beans
Acronym: GIF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Responsible Party: Principal Investigator, JeyaKumar Henry, Principal Investigator, Singapore Institute of Food and Biotechnology Innovation
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2016/00926
Record Dates: First submitted 2019-03-07; First posted 2019-03-11 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2019-03

CONDITIONS: Diabetes Mellitus, Type 2; Obesity; PreDiabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Prediabetic State | interventions — Sucrose

STUDY DESIGN:
Intervention Model Description: Crossover randomized controlled Trials
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Glucose Reference 1 (Other): Glucose solution containing 30 g of glucose
  Interventions: Other: Glucose Reference 1
- Glucose Reference 2 (Other): Glucose solution 2 containing 30 g of glucose
  Interventions: Other: Glucose Reference 2
- Glucose Reference 3 (Other): Glucose solution 3 containing 30 g of glucose
  Interventions: Other: Glucose reference 3
- Sucrose (Experimental): Sucrose solution containing 30 g of sucrose
  Interventions: Other: Sucrose
- Regular Bake beans in tomato sauce (Experimental): Bake bean in tomato sauce with high levels of sucrose (37%)
  Interventions: Other: Regular Bake beans in tomato sauce
- Bake beans in tomato sauce, reduced sugar (Experimental): Bake bean in tomato sauce with medium levels of sucrose (29.9%)
  Interventions: Other: Bake beans in tomato sauce, reduced sugar
- Bake beans in tomato sauce, low GI (Experimental): Bake bean in tomato sauce with low levels of sucrose (18.5%)
  Interventions: Other: Bake beans in tomato sauce, low GI

INTERVENTIONS:
Other: Glucose Reference 1 — 30 g of glucose dissolved in 250 ml of water
  Arms: Glucose Reference 1
Other: Glucose Reference 2 — 30 g of glucose dissolved in 250 ml of water
  Arms: Glucose Reference 2
Other: Glucose reference 3 — 30 g of glucose dissolved in 250 ml of water
  Arms: Glucose Reference 3
Other: Sucrose — 30 g of Sucrose dissolved in 250 ml of water
  Arms: Sucrose
Other: Regular Bake beans in tomato sauce — Bake beans in tomato sauce containing 14 g of sugar
  Arms: Regular Bake beans in tomato sauce
Other: Bake beans in tomato sauce, reduced sugar — Bake beans in tomato sauce containing 12.2 g of sugar
  Arms: Bake beans in tomato sauce, reduced sugar
Other: Bake beans in tomato sauce, low GI — Bake beans in tomato sauce containing 7.2 g of sugar
  Arms: Bake beans in tomato sauce, low GI

SUMMARY:
To investigate the effect of added sugar to bake beans on glycemic and insulinemic response.

DETAILED DESCRIPTION:
There will be a total of 7 test session. Each session will last for 3 hours. At each test session, volunteers will be served with 7 test meals and blood will be collected. After an overnight fast, subjects will visit the research center. Two fasting capillary blood samples will be collected via fingerpick. Following the fasting samples, volunteers will consume the test meals. Further blood samples will be collected at 15, 30, 45, 60, 90, 120, 150, 180 minutes after the ingestion of test meal. These samples will be used to analyses for whole capillary blood glucose. At every 30 minute interval, samples will be collected for analysis of capillary plasma insulin.

ELIGIBILITY:
Inclusion Criteria:

* Chinese ethnicity
* Age ≥21 and ≤ 60 years
* Body mass index between 18.5 to 25 kg/m2
* Normal blood pressure <140/90 mmHg
* Fasting blood glucose <6.0 mmol/L
* In general good health

Exclusion Criteria:

* Current Smoker
* have any metabolic diseases (such as diabetes, hypertension etc)
* have known glucose-6-phosphate dehydrogenase deficiency (G6PD deficiency)
* having medical conditions and/or taking medications known to affect glycaemia (glucocorticoids, thyroid hormones, thiazide diuretics)
* have intolerances or allergies to any foods
* partake in sports at the competitive and/or endurance levels
* intentionally restrict food intake

Ages: 21 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy Male Volunteers
Enrollment: 12 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2019-04-17 (Actual); Study Completion 2019-04-17 (Actual)

PRIMARY OUTCOMES:
Glucose [ | Up to 180 minutes
  Whole capillary blood glucose will be measure using Hemocue analyser

SECONDARY OUTCOMES:
Insulin | Up to 180 minutes
  Capillary plasma will be measure using Cobas analyser

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition Research Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No